CLINICAL TRIAL: NCT00978315
Title: Randomised, Multi-centre, Double-blind, Placebo-controlled Trial of Vitamin D Supplementation in Adult and Adolescent Patients With Asthma
Brief Title: Trial of Vitamin D Supplementation in Asthma
Acronym: ViDiAs
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Barts & The London NHS Trust (Other)
Collaborators: National Health Service, United Kingdom (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 2009-010083-42
Record Dates: First submitted 2009-09-14; First posted 2009-09-16 (Estimated); Last update posted 2014-02-04 (Estimated); Status verified 2014-02

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma | interventions — Cholecalciferol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Vigantol oil (Active Comparator): Vigantol oil will be administered in 2-monthly oral bolus doses over a period of one year
  Interventions: Dietary Supplement: Cholecalciferol
- Miglyol oil (Placebo Comparator): Miglyol oil will be administered in 2-monthly oral bolus doses over a period of one year
  Interventions: Dietary Supplement: Miglyol oil

INTERVENTIONS:
Dietary Supplement: Cholecalciferol — Cholecalciferol will be administered as 2-monthly oral bolus doses of Vigantol oil over a period of one year
  Arms: Vigantol oil
Dietary Supplement: Miglyol oil — Miglyol oil will be administered as 2-monthly oral bolus doses of Vigantol oil over a period of one year
  Arms: Miglyol oil

SUMMARY:
The study null hypothesis is that vitamin D supplementation will not influence time to upper respiratory tract infection or time to severe asthma exacerbation in adult and adolescent patients with asthma.

ELIGIBILITY:
Principal Inclusion Criteria:

* Medical record diagnosis of asthma
* Age ≥ 16 years and ≤ 80 years on day of first dose of IMP
* If a woman of child-bearing potential, is sexually abstinent or has negative pregnancy test within 7 days of recruitment and agrees to use reliable form of contraception until she has completed the study
* Able to give written informed consent to participate in the study

Principal Exclusion Criteria:

* Diagnosis of COPD
* Known sarcoidosis, hyperparathyroidism, nephrolithiasis, active tuberculosis, vitamin D intolerance, liver failure, renal failure, terminal illness, lymphoma or other malignancy not in remission for ≥ 3 years
* Any other condition that, in an investigator's judgement, might compromise patient safety or compliance, interfere with evaluation or preclude completion of the study
* Taking benzothiadiazine derivative, cardiac glycoside, carbamazepine, phenobarbital, phenytoin or primidone
* Taking dietary supplement containing vitamin D up to 2 months before first dose of IMP
* Treatment with any investigational medical product or device up to 4 months before first dose of IMP
* Breastfeeding, pregnant or planning a pregnancy
* Baseline corrected serum calcium > 2.65 mmol/L
* Baseline serum creatinine > 125 micromol/L
* Smoking history >15 pack-years

Ages: 16 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 250 (Actual)
Dates: Start 2009-09; Primary Completion 2013-07 (Actual); Study Completion 2013-07 (Actual)

PRIMARY OUTCOMES:
Time to first upper respiratory tract infection | One year
Time to first severe asthma exacerbation | One year

SECONDARY OUTCOMES:
Asthma Control Test Score | One year
Time to unscheduled health service use for upper respiratory tract infection or severe asthma exacerbation | One year
Proportion of participants experiencing hypercalcaemia | One year

CONTACTS AND LOCATIONS:
Overall Officials: Adrian R Martineau, MRCP, Study Director — Queen Mary University of London
Locations (4):
- United Kingdom (4):
  - Barts and The London NHS Trust, London, London
  - Lower Clapton Health Centre, London, London
  - Homerton University Hospital NHS Foundation Trust, London, London
  - Guy's and St Thomas' NHS Foundation Trust, London, London

REFERENCES:
- [Derived] Martineau AR, MacLaughlin BD, Hooper RL, Barnes NC, Jolliffe DA, Greiller CL, Kilpin K, McLaughlin D, Fletcher G, Mein CA, Hoti M, Walton R, Grigg J, Timms PM, Rajakulasingam RK, Bhowmik A, Rowe M, Venton TR, Choudhury AB, Simcock DE, Sadique Z, Monteiro WR, Corrigan CJ, Hawrylowicz CM, Griffiths CJ. Double-blind randomised placebo-controlled trial of bolus-dose vitamin D3 supplementation in adults with asthma (ViDiAs). Thorax. 2015 May;70(5):451-7. doi: 10.1136/thoraxjnl-2014-206449. Epub 2015 Feb 27. PMID 25724847